CLINICAL TRIAL: NCT02448004
Title: A Phase 1, Open-label Study to Characterize the Absorption, Metabolism and Excretion of 14C-JNJ-63623872 After a Single Dose in Healthy Male Subjects
Brief Title: Study to Assess the Absorption, Metabolism and Excretion of 14C-JNJ-63623872 After a Single Dose in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107301; 63623872FLZ1007 (Other: Janssen Cilag N.V./S.A., Belgium); 2015-000719-42 (EudraCT Number)
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Healthy; JNJ-63623872; 14C-JNJ-63623872
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- JNJ-63623872 (Experimental): Participants will receive a single 600-milligram (mg) dose of JNJ-63623872 administered as three capsules containing 14C-labeled and unlabeled JNJ-63623872.
  Interventions: Drug: JNJ-63623872

INTERVENTIONS:
Drug: JNJ-63623872 — Participants will receive a single 600-mg dose of JNJ-63623872 administered as three capsules containing 14C-labeled and unlabeled JNJ-63623872.
  Other Names: 14C-JNJ-63623872

SUMMARY:
The primary objective of this study is to characterize the absorption and metabolic pathways of JNJ-63623872, and the excretion of the compound and its metabolites, after single oral dosing of 14C-JNJ-63623872 in healthy adult male participants.

DETAILED DESCRIPTION:
This is a Phase 1, open-label (all people know the identity of the intervention), single dose study in 6 healthy adult male participants to characterize the absorption, metabolism and excretion of 14C-JNJ-63623872. The total study duration will be approximately of 16 days per participant. The study consists of 3 parts: Screening (that is, 28 days before study commences on Day 1); open-Label Treatment Phase(that is, Day 1); and Follow-up (that is, up to Day 16). All the eligible participants will receive 14C-JNJ-63623872 at a dose level of 600 milligram. Participants will enter the study site on Day -1 and stay at the study site at least until Day 8. Urine, feces, whole blood samples, plasma, nasal mucus and saliva samples will be collected up to Day 8. Unchanged JNJ-63623872 will be determined in plasma and, if feasible, in saliva. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must agree to comply with contraceptive measures as mentioned in protocol
* Must be non-smokers for at least 3 months prior to screening
* Must have a Body Mass Index (BMI; weight in kilogram divided by the square of height in meters) of 18.0 to 30.0 kilogram/meter square, extremes included
* Must have signed an Informed consent form indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study before starting any screening activities
* Must be willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Must have a normal 12-lead ECG (based on the mean value of the triplicate parameters) at screening and on Day 1 predose including: 1). normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); 2). QT interval corrected for heart rate according to Fridericia (QTcF) interval less than or equal to (<=) 450 milliseconds (ms); 3). QRS interval lower than 120 ms; 4). PR interval <= 220 ms

Exclusion Criteria:

* Participants with a past history of heart arrhythmias (extrasystoli clinically significant in the opinion of the investigator, tachycardia at rest) or of risk factors for Torsade de Pointes syndrome
* Participants with more than one episode of constipation (less than 1 stool per 3 days) during the last 2 months, or more than one episode of diarrhea (3 or more stools per day) during the last 2 months
* Participants with a history of or a reason to believe the subject has a history of drug or alcohol abuse within the past 5 years
* Participants having a positive urine drug test at study screening or on Day -1. Urine will be tested for the presence of amphetamines, benzodiazepines, cocaine, cannabinoids, opioids, methadone and barbiturates
* Participants with documented human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection at study screening
* Participants with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M ([IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen [HbsAg]), or hepatitis C virus (HCV) infection (confirmed by HCV antibody) at study screening

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2015-06-24 (Actual); Study Completion 2015-06-24 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-63623872 | Baseline up to Day 8
  The Cmax is the maximum plasma concentration.
Time to reach maximum concentration (tmax) of JNJ-63623872 | Baseline up to Day 8
  The Tmax is time to reach the maximum plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last (AUC [0-last]) of JNJ-63623872 | Baseline up to Day 8
  AUC from time 0 to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-63623872 | Baseline up to Day 8
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Terminal Half-Life(t[1/2]) of JNJ-63623872 | Baseline up to Day 8
  Terminal half-life (t[(1/2]) is defined as 0.693/Lambda(z).
Rate Constant (Lambda[z]) | Baseline up to Day 8
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent total body clearance (CL/F) of JNJ-63623872 | Baseline up to Day 8
  Clearance is a quantitative measure of the rate at which a drug substance is removed from the body. The CL/F will be calculated by dividing the dose by AUC (0-infinity).
Apparent volume of distribution at the terminal Phase (Vd[z] /F) of JNJ-63623872 | Baseline up to Day 8
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.The Vd(z)/F will be calculated by dividing CL/F by lambda(z).
Amount of JNJ-63623872 excreted in Urine (Ae[x-y]) | Baseline up to Day 8
  Amount excreted into urine over a given time interval, calculated from the urinary drug concentration of the collection interval x to y hours post dosing multiplied with the associated urine volume of the interval.
Total Amount of JNJ-63623872 excreted in Urine (Ae[total]) | Baseline up to Day 8
  Total amount excreted into urine, calculated by adding the amounts of the individual intervals together.
Percentage of JNJ-63623872 dose excreted into urine | Baseline up to Day 8
  Percentage of the dose excreted into urine of the collection interval x to y hours post dosing, calculated as 100 x (Aex-y/Dose).
Total Percentage of JNJ-63623872 dose excreted into urine | Baseline up to Day 8
  Total percentage of the dose excreted into urine, calculated as 100 * (Ae[total]/Dose).
Renal clearance | Baseline up to Day 8
  Renal clearance calculated as Ae (total)/AUC (infinity).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.
Locations (1):
- Groningen, Netherlands